CLINICAL TRIAL: NCT07341009
Title: Evaluation of a Neuropsychological Tool to Assess Temporal Processing Abilities in Alzheimer's Disease
Acronym: CHRONOS
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 25-0136
Record Dates: First submitted 2025-12-12; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-10

CONDITIONS: Alzheimer's Disease (AD); Time Perception
Keywords: temporal cognition; dementia; cognition; neuropsychology
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Alzheimer's patients
  Interventions: Behavioral: Chronos battery

INTERVENTIONS:
Behavioral: Chronos battery — Patients will perform the battery during a neuropsychological assessment

SUMMARY:
Perceiving and representing the passage of time allows us to temporally organize perceptions and memories for the coordination of actions, planning, and the mobilization of cognitive processes toward a goal. This innovative project aims to clarify the profile of time impairment associated with normal aging and the progression of age-related pathologies. This project proposes to develop a new neuropsychological tool for quantifying and preventing changes in the relationship to time associated with Alzheimer's disease. Four aspects of time are distinguished, which are measured separately and distributed along a continuum between perception and memory: (a) perception of simultaneity and order; (b) processing of durations; (c) subjective sense of the passage of time; and (d) mental time travel. Crucially, many neurological and psychiatric disorders are associated with impairment in one or more aspects of time. However, time remains largely unexplored in clinical practice. Patients with Alzheimer's disease will complete the CHRONOS battery. This battery allows for a rapid assessment (approximately ten minutes) of the four aspects of time. This new battery will enable the identification of behavioral markers aimed at improving prognosis and prevention regarding individual cognitive trajectories of aging. The relationship to time is closely linked to each person's personal experience. This project will help to put into words difficulties that are not always expressed in terms of time. Thus, considering these pathologies from the perspective of time aims to better understand and prevent their difficulties and to guide the identification of new markers and new avenues for remediation.

ELIGIBILITY:
Inclusion Criteria:

* No objection from the participant or their legal representative, if applicable, prior to or during the assessment
* Deficit in at least two cognitive functions, including episodic memory.

Exclusion Criteria:

* History of head trauma with loss of consciousness lasting more than 1 hour
* Presence of clinically significant major psychiatric disorders (according to DSM-IV-TR criteria)
* Use of medications likely to alter cognitive and/or brain function (decision by the principal investigator)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Alzheimer's disease
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Behavioral difference at the battery assessing temporal processing (CHRONOS Score) | From enrollment to the end of the neuropsychological assessment (three hours)

CONTACTS AND LOCATIONS:
Locations (1):
- Caen Hospital, neurology Unit, Caen, France

IPD SHARING:
Plan to Share IPD: No